CLINICAL TRIAL: NCT02995525
Title: Prevalence of Chronic Pain After Scoliosis and Thoracic Surgery in Children
Brief Title: Chronic Pain After Scoliosis and Thoracic Surgery in Children
Acronym: PEDIACHROII
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBXSAR32016-02
Record Dates: First submitted 2016-11-10; First posted 2016-12-16 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2016-12

CONDITIONS: Thoracic Surgery; Scoliosis; Adolescence; Pediatric ALL; Chronic Pain
MeSH Terms: conditions — Scoliosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this epidemiologic prospective study is to determine the prevalence of CPSP defined as pain occurring 4 months after scoliosis and thoracic surgery and rated > 3 on a 10 point visual analogue scale or FLACC scale, in children aged from 6 to 18 years.

The main objective : prevalence of chronic post surgical pain 4 months after scoliosis ant thoracic surgery in children aged 6 to 18 years.

The secondary objectives: the intensity of chronic post surgical pain, the prevalence of neuropathic syndrome and the predictive risk factors.

ELIGIBILITY:
Inclusion Criteria:

* children aged from 6 to 18 years undergoing scoliosis or thoracic surgery in paediatric Bordeaux hospital.

Exclusion Criteria:

* patients who not willing to participate, with children and/or parental insufficient understanding of the questionnaires.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children aged from 6 to 18 years undergoing scoliosis or thoracic surgery in paediatric Bordeaux hospital
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
pain at 4 months after surgery | 4 months after scoliosis and thoracic surgery in children aged 6 to 18 years
  visual analogue scale for pain (0_100)

SECONDARY OUTCOMES:
adverse events after surgery | adverse events during peri-operative period (hospital stay, i.e. during the first month after surgery)
  infections, neurologic defect, new surgery, blood hematoma
morphine consumption during the perioperative period | the perioperative period (preoperative period i.e. more than 1 month before, the month before, the before surgery; during hospitalization)
  morphine consumption (mg/day)
pain during the perioperative period | the perioperative period (preoperative period i.e. more than 1 month before, the month before, the before surgery; during hospitalization)
  visual analogue scale for pain (0-100)
pain during the perioperative period in disabled children aged 6 to 18 years | the perioperative period (preoperative period i.e. more than 1 month before, the month before, the before surgery; during hospitalization)
  FLACC scale level (0-100)
prevalence of neuropathic syndrome during perioperative period and at 4 months after surgery | 2'4-48 h hours period after surgery, 4 months after surgery
  DN4 questionnaire
pain at 4 months after surgery | 4 months after scoliosis and thoracic surgery in disabled children aged 6 to 18 years
  modified FLACC scale for pain

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier Universitaire de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Batoz H, Semjen F, Bordes-Demolis M, Benard A, Nouette-Gaulain K. Chronic postsurgical pain in children: prevalence and risk factors. A prospective observational study. Br J Anaesth. 2016 Oct;117(4):489-496. doi: 10.1093/bja/aew260. Epub 2016 Oct 17. PMID 28077537